CLINICAL TRIAL: NCT06030466
Title: A Comparative Study of Medical Students' Acceptance and Learning Efficacy With Physical and Virtual Standardized Patients
Brief Title: Medical Students' Acceptance and Learning Efficacy With Physical and Virtual Standardized Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202307039RINA
Record Dates: First submitted 2023-08-24; First posted 2023-09-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Education, Medical

STUDY DESIGN:
Intervention Model Description: Randomization with crossover design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With physical standardized patients (Other): Medical students practice consultation with physical standardized patients.
  Interventions: Other: With physical standardized patients
- With virtual standardized patients (Experimental): Medical students practice consultation with virtual standardized patients.
  Interventions: Other: With virtual standardized patients

INTERVENTIONS:
Other: With virtual standardized patients — The virtual standardized patient is a software system that presents on a computer screen like a video conference, allowing medical students to interact with it for medical consultation. The virtual character modeling adopts 3D model, the expression of the character is delicate, and the voice feedback is clear. After the students' questions are asked by voice recognition and key words are extracted, appropriate responses are given.
  Arms: With virtual standardized patients
Other: With physical standardized patients — The physical standardized patient is a real person who has received professional training courses in the department of medical education of National Taiwan University Hospital, and can help medical students practice consultations.
  Arms: With physical standardized patients

SUMMARY:
This study will focus on exploring the experiential differences between virtual standardized patients and physical standardized patients, gathering feedback through questionnaires and brief interviews. Standardized patients have been widely used in medical education and physician licensing exams in Taiwan for over 15 years. With the rise of technology-enhanced medical education, it is necessary to reexamine the professional attributes and identification of standardized patients and explore the implementation of virtual standardized patient systems. The research aims to reshape the professional identity of standardized patients, identify necessary attributes and competencies, and establish a virtual standardized patient system to assess medical students' acceptance and learning outcomes.

DETAILED DESCRIPTION:
This research project aims to investigate the differences in acceptance and learning efficacy between physical standardized patients and virtual standardized patients among medical students. Participants will be randomly assigned to either the physical standardized patient group or the virtual standardized patient group. They will experience scenarios with real standardized patients or screen-based virtual standardized patients, engaging in activities such as taking medical histories and explaining conditions. The study will collect questionnaire feedback on learning efficacy and acceptance.

The primary research questions include: Are there differences in medical students' perceptions of teaching scenarios involving virtual standardized patients versus physical standardized patients? Are there differences in medical students' self-efficacy growth after practicing teaching scenarios with virtual standardized patients versus real standardized patients? Secondary research questions include: What professional attributes and competencies should standardized patients possess? Does technological literacy influence medical students' acceptance of virtual standardized patients? How do virtual and physical standardized patient scenarios differ in terms of perceptions by standardized patients and learners?

This study will focus on exploring the experiential differences between virtual standardized patients and physical standardized patients, gathering feedback through questionnaires and brief interviews. Standardized patients have been widely used in medical education and physician licensing exams in Taiwan for over 15 years. With the rise of technology-enhanced medical education, it is necessary to reexamine the professional attributes and identification of standardized patients and explore the implementation of virtual standardized patient systems. The research aims to reshape the professional identity of standardized patients, identify necessary attributes and competencies, and establish a virtual standardized patient system to assess medical students' acceptance and learning outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Medical students studying at the National Taiwan University School of Medicine
2. Able to understand the research case and sign the written consent form

Exclusion Criteria:

1. Has used relevant virtual standardized patient software in the past (past exposure)
2. Unable to adapt to technological applications or successfully use this virtual standardized patient system (unable to cooperate with research)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Perception differences between medical student using virtual standardized patients and physical standardized patients. | 1 year
  Perception questionnaire including satisfaction and acceptability. The questionnaire will use a 5-Point Likert Scale to assess the acceptance and satisfaction levels of physical standardized patients in comparison to virtual standardized patients among medical students. Here are some sample questions:
  S1: I am satisfied with how the "Virtual Standardized Patient System" operates.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  S2: I am satisfied with the interactive process of medical history inquiries within the "Virtual Standardized Patient System."
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  S3: I am satisfied with the interactive process of medical condition explanations within the "Virtual Standardized Patient System."
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Learning efficacy difference between medical student using virtual standardized patients and physical standardized patients. | 1 year
  The questionnaire will employ a 5-Point Likert Scale to investigate the learning effectiveness of medical students when comparing physical and virtual standardized patients. Below are some sample questions:
  PU2: I believe that the "Virtual Standardized Patient System" can be expected to enhance clinical learning.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  PU3: I am of the opinion that the "Virtual Standardized Patient System" will facilitate clinical learning.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  EE4: I find learning to use the "Virtual Standardized Patient System" to be a challenging skill to master.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Heng Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Medical Education, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No